CLINICAL TRIAL: NCT06318585
Title: Creazione di un Database Clinico Per lo Studio Della variabilità Fenotipica Nella Malattia Del Motoneurone
Brief Title: Creation of a Clinical Database for the Study of Phenotypic Variability in Motor Neuron Diseases
Acronym: ALS-PHENO
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C306
Record Dates: First submitted 2024-03-08; First posted 2024-03-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma, serum, CSF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Description: Characterization of Motor Neuron Disease Phenotypes

The goal of this observational study is to understand the clinical presentation of motor neuron disease (MND) in patients attending the Neurology Department of the Istituto Auxologico Italiano. The main questions it aims to answer are:

* What are the specific clinical phenotypes associated with MND?
* How can these phenotypes contribute to a better understanding of the disease's underlying mechanisms and improve prognostic accuracy?

Participants will undergo:

* Clinical evaluation using validated scales
* Neurophysiological and neuroradiological instrumental assessment
* Neuropsychological evaluation
* Collection of biological materials for genetic screening and biomarker assessment, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ALS or other motor neuron disease

Exclusion Criteria:

* refusal to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cohort of patients from a tertiary Italian ALS Centre
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
no. of patients with classic ALS | baseline (at diagnosis), at 1 year
  no. of patients with classic ALS
no. of patients with bulbar ALS | baseline (at diagnosis), at 1 year
  no. of patients with bulbar ALS
no. of patients with LMN phenotypes (flail arm, flail leg, PMA) | baseline (at diagnosis), at 1 year
  no. of patients with LMN phenotypes (flail arm, flail leg, PMA)
no. of patients with UMN phenotypes (pyramidal ALS, PLS) | baseline (at diagnosis), at 1 year
  no. of patients with UMN phenotypes (pyramidal ALS, PLS)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luca, Milan, MI, Italy